CLINICAL TRIAL: NCT01920958
Title: Use of Tachosil® for Lymph Sealing During Surgery. A Non-Interventional Study
Brief Title: Use of Tachosil® for Lymph Sealing During Surgery
Acronym: SEAL
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TC-2402-401-DE; U1111-1142-0279 (Registry Identifier: WHO)
Record Dates: First submitted 2013-07-19; First posted 2013-08-12 (Estimated); Results first posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-10

CONDITIONS: Lymph Node Resection
MeSH Terms: interventions — TachoSil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TachoSil®: TachoSil®, sterile absorbable patch, topical application, used during surgery in participants who had lymphadenectomy according to the Summary of Product Characteristics.
  Interventions: Other: TachoSil®

INTERVENTIONS:
Other: TachoSil® — TachoSil® is a collagen sponge that is coated with the active substances human fibrinogen and human thrombin and that supports hemostasis and tissue sealing in surgery.

SUMMARY:
The purpose of this study is to describe effectiveness and reliability of TachoSil® in lymph sealing after lymphadenectomy.

DETAILED DESCRIPTION:
The aim of this non-interventional study (NIS) was to collect further knowledge on the routine use of TachoSil ® in lymph node surgery where its sealing property helps to reduce the rate of postoperative complications, especially of seroma formation. Some data are already available from gynecology, urology and thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Stationary patients undergoing lymph node resection.

Exclusion Criteria:

* Contraindications, such as hypersensitivity to the active pharmaceutical ingredient or to another ingredient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stationary patients in whom a lymph node resection was planned to be performed
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2012-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda Pharma Vertrieb GmbH & Co. KG
Locations (1):
- Greifswald, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 39 investigative sites in Germany from 30 September 2012 to 27 March 2014.
Pre-assignment Details: Collection of information of routine use of TachoSil® in participants who had lymph node surgery.
Groups:
- TachoSil®: TachoSil®, sterile absorbable patch, topical application, applied during surgery in participants who had lymph node surgery according to the Summary of Product Characteristics.
Period: Overall Study
Arm/Group | TachoSil®
Started | 233
Completed | 228 (Intent-to-Treat (ITT) Population)
Not Completed | 5
Not completed — Did Not Fulfill Inclusion Criteria | 5

BASELINE CHARACTERISTICS:
Population: ITT population consisted of all patients who received patient information and who consented to the collection, transmission and evaluation of their data and who underwent lymph node resection with TachoSil®.
Arm/Group | TachoSil®
Number analyzed (Participants) | 228
Age, Continuous [Mean (Standard Deviation); unit: years] — Age data was available for 226 participants.
  years | 63.6 (10.82)
Sex/Gender, Customized [Number; unit: participants]
  Female | 110
  Male | 111
  Missing | 7
Region of Enrollment [Number; unit: participants]
  Germany | 228
Height [Mean (Standard Deviation); unit: cm] — Height data was available for 216 participants.
  cm | 169.9 (9.07)
Weight [Mean (Standard Deviation); unit: kg] — Weight data was available for 216 participants.
  kg | 79.6 (15.84)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI data was available for 216 participants.
  kg/m^2 | 27.55 (5.092)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Post-Operative Seroma Formation Over Time as Determined at Hospital Discharge
Time Frame: Up to 50 Days
Population: Intent-to-treat population consisted of all participants who received patient information, signed consent and had Tachosil® applied during lymph node surgery.
Measure: Number; unit: percentage of participants
Arm/Group | TachoSil®
Number analyzed (Participants) | 228
percentage of participants | 2.63

2. Secondary Outcome: Assessment of TachoSil® by the Surgeon With Respect to Handling Using a 10-Point Numerical Rating Scale
Description: The surgeon evaluated handling of TachoSil® using a 10-point scale where: 1=very good to 10=very poor.
Time Frame: Peri- and post-surgery (Up to 50 Days)
Population: Participants from the Intent-to-treat population (all participants who received patient information, signed consent and had Tachosil® applied during lymph node surgery) with data available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TachoSil®
Number analyzed (Participants) | 225
score on a scale | 2.2 (0.98)

3. Secondary Outcome: Assessment of TachoSil® by the Surgeon With Respect to Utility in Operation Using a 10-Point Numerical Rating Scale
Description: The surgeon evaluated Utility in Operation of TachoSil® using a 10-point scale where: 1=very useful to 10=completely useless.
Time Frame: Peri- and post-surgery (Up to 50 Days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TachoSil®
Number analyzed (Participants) | 225
score on a scale | 2.3 (1.25)

4. Secondary Outcome: Assessment of TachoSil® by the Surgeon With Respect to Satisfaction Using a 10-Point Numerical Rating Scale
Description: The surgeon evaluated Satisfaction in Operation of TachoSil® using a 10-point scale where: 1=very satisfied to 10=totally unsatisfied.
Time Frame: Peri- and post-surgery (Up to 50 Days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TachoSil®
Number analyzed (Participants) | 225
score on a scale | 2.3 (1.42)

5. Secondary Outcome: Percentage of Participants With at Least One Drainage Inserted
Description: The total number of participants where at least one drainage was used during the operation.
Time Frame: Baseline (Day of Surgery)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | TachoSil®
Number analyzed (Participants) | 228
percentage of participants | 81.14

6. Secondary Outcome: Percentage of Participants With Change in Length of Drainage Stay and Drainage Volume
Time Frame: Up to 50 Days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | TachoSil®
Number analyzed (Participants) | 185
percentage of participants
  Change in Length of Drainage Stay | 48.65
  Change in Drainage Volume | 57.84

7. Secondary Outcome: Length of Hospital and ICU Stay
Description: Length of stay includes time (days) spent in the intensive care unit (ICU) and normal hospital station.
Time Frame: Up to 50 Days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TachoSil®
Number analyzed (Participants) | 228
days
  Hospital Stay (n=225) | 12.2 (6.57)
  ICU Stay (n=100) | 2.8 (1.91)

8. Secondary Outcome: Percentage of Participants With Pharmacoeconomic Benefit Based on Savings of Operating Time
Description: Pharmacoeconomic benefit was assessed by the surgeon based on savings/shortening of operating time in minutes.
Time Frame: Peri- and post-surgery (Up to 50 Days)
Population: ITT population consisted of all patients who received patient information and consented to the collection, transmission and evaluation of their data and who underwent lymph node resection with TachoSil®.
Measure: Number; unit: percentage of participants
Arm/Group | TachoSil®
Number analyzed (Participants) | 228
percentage of participants | 17.98

9. Secondary Outcome: Percentage of Participants With Pharmacoeconomic Benefit Based on Shortening of Hospital Stay
Description: Pharmacoeconomic benefit was assessed by the surgeon at hospital discharge based on shortening of hospital stay in days.
Time Frame: Up to 50 Days
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | TachoSil®
Number analyzed (Participants) | 228
percentage of participants | 27.19

10. Secondary Outcome: Percentage of Participants With Pharmacoeconomic Benefit in Shortening of Time Spent in ICU
Description: Pharmacoeconomic benefit was assessed by the surgeon at hospital discharge based on shortening of time spent in ICU in days.
Time Frame: Up to 50 Days
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | TachoSil®
Number analyzed (Participants) | 228
percentage of participants | 8.77

11. Secondary Outcome: Percentage of Participants With Pharmacoeconomic Benefit Based on Drainage Time Reduced
Description: Pharmacoeconomic evaluation as assessed by the surgeon at hospital discharge based on drainage time reduced in days.
Time Frame: Up to 50 Days
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | TachoSil®
Number analyzed (Participants) | 228
percentage of participants | 35.96

12. Secondary Outcome: Percentage of Participants With Pharmacoeconomic Benefit Based on Drainage Volume Reduced
Description: Pharmacoeconomic benefit was assessed by the surgeon at hospital discharge based on the drainage volume reduced in milliliters.
Time Frame: Up to 50 Days
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | TachoSil®
Number analyzed (Participants) | 228
percentage of participants | 39.04

13. Secondary Outcome: Percentage of Participants With Post-Operative Complications and Adverse Events
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Up to 50 Days
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | TachoSil®
Number analyzed (Participants) | 228
percentage of participants
  Postoperative Complications | 18.42
  Adverse Events | 13.60

ADVERSE EVENTS:
Time Frame: Up to 30 days
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TachoSil®
Serious Adverse Events (participants affected / at risk) | 7/228
Other Adverse Events (participants affected / at risk) | 25/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TachoSil® (N=228)
Groin abscess (Infections and infestations) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2
Seroma (Injury, poisoning and procedural complications) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Lymphocele (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TachoSil® (N=228)
Lymphocele (Vascular disorders) | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.